CLINICAL TRIAL: NCT04041063
Title: Rehabilitation and Cortical Remodeling After Surgical Intervention for Spinal Cord Injury
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Burke Medical Research Institute (Other)
Collaborators: Massachusetts General Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: SCI_nerve_transfer_robotics
Record Dates: First submitted 2019-07-30; First posted 2019-08-01 (Actual); Last update posted 2024-08-23 (Actual); Status verified 2024-08

CONDITIONS: Spinal Cord Injuries; Tetraplegia; Cervical Spinal Cord Injury
Keywords: robotics, hand function
MeSH Terms: conditions — Spinal Cord Injuries; Quadriplegia

STUDY DESIGN:
Intervention Model Description: All participants will receive nerve transfer surgery. Half of the participants will receive 6 weeks of robotic training starting one year after the surgery. The other half of the participants will receive 6 weeks of robotic training starting one year plus 6 weeks after the nerve transfer surgery.
Who Masked: Outcomes Assessor
Masking Description: The outcomes assessor will not have knowledge of the time point at which they are assessing the participant.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Nerve transfer + robotic training (Experimental): Participants will receive nerve transfer surgery at Massachusetts General Hospital in Boston, MA. One year after the surgery, participants will receive six weeks of upper limb robotic training at the Burke Neurological Institute in White Plains, NY.
  Interventions: Device: Upper limb robotic training; Procedure: Nerve transfer surgery
- Nerve transfer + delayed robotic training (Active Comparator): Participants will receive nerve transfer surgery at Massachusetts General Hospital in Boston, MA. One year + six weeks after the surgery, participants will receive six weeks of upper limb robotic training at the Burke Neurological Institute in White Plains, NY.
  Interventions: Device: Upper limb robotic training; Procedure: Nerve transfer surgery

INTERVENTIONS:
Device: Upper limb robotic training — Subjects will remain seated in their own wheelchair in front of the InMotion Hand™ Robot (Interactive Motion Technologies, Massachusetts, MA, Figure 6) facing a video screen.
  The arm of the participants will be abducted, forearm supported, and hand grasping a cone shaped handle. Velcro straps will lightly hold the forearm and fingers secure. The InMotion Hand™ robot attaches to the InMotion Arm™ robots to provide 'assisted-as-needed'™ gross grasp and release motion and support for functional reach. In each session, patients perform a total of 1024 movement repetitions (Cortes et al., 2013). Patients will receive a total of 18 sessions (3x/week, 6 weeks) comprising one hour of interactive hand robotic training. The interactive robotic features involve visuomotor task, moving the robotic manipulandum according to targets on a computer screen mounted at eye level.
Procedure: Nerve transfer surgery — C5 injury; Teres minor branch of axillary nerve transferred to long head of triceps branch of radial nerve (RN); Brachialis branch of musculocutaneous nerve to anterior interosseous nerve (AIN); Supinator branch of RN to posterior interosseous nerve (PIN). C6 injury; Teres minor branch of axillary nerve to long head of triceps branch of RN; Extensor carpi radialis brevis (ECRB) branch of RN to AIN; Supinator branch of RN to PIN. C7 injury with preserved triceps, loss of grasp/release; Pronator teres branch of median nerve to AIN; Terminal branch of ECRB branch of RN to flexor pollicis longus branch of AIN; Supinator branch of RN transferred to PIN. C7 injury with preserved triceps/finger extension, loss of grasp; Pronator teres branch of median nerve to AIN; Terminal branch of ECRB branch of RN to flexor pollicis longus branch of AIN.

SUMMARY:
The aim of this study is to determine the effects of rehabilitation on dexterous hand movements and cortical motor map changes in tetraplegic patients following nerve transfer surgery. The working hypothesis is that robot-assisted, intensive rehabilitation will support the return of hand and arm function and strengthen the cortical representations of targeted muscles. The investigators will assess this through TMS mapping and clinical measures of hand and arm function.

DETAILED DESCRIPTION:
The recovery of hand and arm function is of critical importance for decreasing long-term care costs and increasing quality of life for individuals with tetraplegia due to spinal cord injury (SCI). A subset of these individuals, with injuries in the mid to low cervical spinal cord, are candidates for nerve transfer surgery. Nerve transfer surgery restores function after SCI through coaptation of redundant, intact donor nerves to recipient nerves arising at or below the level of SCI. The use of nerve transfer after SCI is relatively novel and many patients exhibit a remarkable recovery of hand and arm motor function in the months that follow, however others show a much more limited recovery. The extent of recovery is likely limited, in part, by variability in rehabilitation and the ability of the motor cortex to incorporate the new peripheral circuitry resulting from this surgical procedure. There is a critical need to determine the response of cortical motor networks to nerve transfer and the role that rehabilitation plays in supporting cortical plasticity and motor recovery. If this need is not met, incomplete recovery from this state-of-the-art surgical intervention will persist and the potential application to a wider patient population will not be realized.

The investigators will test the central hypothesis that nerve transfer surgery after cervical SCI creates a novel cortical motor network, which can support the return of dexterous hand/forelimb function through rehabilitation-dependent remodeling. The hypothesis has been based upon 1) previous work in an animal model showing that rehabilitation reshapes cortical motor maps, 2) the pioneering work of a handful of clinicians, including the study collaborator, Justin Brown, that have applied nerve transfer to bypass spinal levels affected by injury, and 3) recent work using transcranial magnetic stimulation (TMS) in human SCI to map the cortical representation of arm muscles in the zone of partial preservation, and the ability to improve hand-arm function through intensive robotic training in chronically impaired subjects. The use of TMS to map cortical motor networks will allow the investigators to measure the cortical reorganization resulting from nerve transfer and determine the extent to which rehabilitation can engage this alternative cortical motor network. The rationale for the proposed studies is that a determination of the mechanisms that support rehabilitation-mediated recovery after nerve transfer will be required for optimizing and refining current clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Tetraplegia (cervical lesion) with some degree of motor dysfunction in the hand
* Motor incomplete or complete lesion (measured by the ASIA Impairment Scale, A, B, C, D).
* Chronic lesion (at least 6months after the injury)
* Demonstrate stability of motor examination for at least six months.
* Retain intact innervation within paralyzed target muscles (axon recipient) as determined by electrodiagnostics.
* Have muscles innervated by the nerves to be used for the transfers (axon donors) of MRC grade 4/5 or greater and sufficient innervation as determined by electrodiagnostics.
* Have access to an at home caregiver who can assist with customary postsurgical physical therapy.
* Ability to give informed consent and understand the tasks involved.

Exclusion Criteria:

* Presence of potential risk factor for brain stimulation: history of seizures, presence of surgically implanted foreign bodies such as a pacemaker, metal plate in the skull, and metal inside the skull.
* History of head trauma and/or cognitive deficit
* Medically unstable
* Contraindicated for nerve transfer surgery.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 6 (Actual)
Dates: Start 2019-07-26 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in Box and Blocks test score | 1 year post surgery, immediately post training, minus baseline before surgery
  The Box and Blocks test measures how many blocks a person can grasp and transfer in one minute. A higher score is associated with better hand function.

SECONDARY OUTCOMES:
Upper extremity motor score (UEMS) | 1 year post surgery, immediately post training, minus baseline before surgery
  The Upper extremity motor score (UEMS) tests the clinical motor strength from 0 to 5 from each key muscle using the ASIA scale. This sum score ranges from 0 (paralyzed) to 25 (normal) in each limb.
Spinal Cord Independence Measure (SCIM III) | 1 year post surgery, immediately post training, minus baseline before surgery
  The Spinal Cord Independence Measure (SCIM III) measures the ability of patients with SCI to perform everyday tasks according to their value for the patient. SCIM is used for quantitative functional outcome assessment following interventions designed to promote recovery from spinal cord injury and to increase functional achievement; and it covers 19 tasks in 16 categories (score range 0-100); all activities of daily living, grouped into four areas of function (subscales): Self-Care (scored 0-20), Respiration and Sphincter Management (0-40), Mobility in Room and Toilet (0-10), Mobility Indoors and Outdoors (0-30).
Modified Ashworth Scale | 1 year post surgery, immediately post training, minus baseline before surgery
  The Modified Ashworth Scale (MAS) will be used to measure change in spasticity. The scale is a scale from 0 to 4 that measures muscle stiffness. A higher score is associated with greater spasticity.
Single pulse transcranial magnetic stimulation | 1 year post surgery, immediately post training, minus baseline before surgery
  Changes in resting motor threshold (RMT), motor evoked potential (MEP) amplitude will be measured in each muscle of both arms using a MagStim X100 stimulator (MagStim) and a figure-8 coil. We will investigate the neurophysiological correlates of function, and the characteristics of participants who respond better to the training.

CONTACTS AND LOCATIONS:
Locations (1):
- Burke Neurological Institute, White Plains, New York, United States

IPD SHARING:
Plan to Share IPD: No